CLINICAL TRIAL: NCT00671970
Title: Phase II Trial of Bevacizumab Plus Erlotinib for Patients With Recurrent Malignant Glioma
Brief Title: Phase (Ph) II Bevacizumab + Erlotinib for Patients (Pts) With Recurrent Malignant Glioma (MG)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000220
Record Dates: First submitted 2008-01-29; First posted 2008-05-06 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-03

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: Glioblastoma; Gliosarcoma; Recurrent MG; Malignant glioma; Glioma; Glioblastoma multiforme (GBM); GBM; Brain tumor; Anaplastic astrocytoma; Anaplastic oligodendroglioma; Anaplastic oligoastrocytoma; Bevacizumab; Avastin; Erlotinib; Tarceva
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms; Astrocytoma; Oligodendroglioma | interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab + Erlotinib (Experimental): Bevacizumab + Erlotinib
  Interventions: Drug: Bevacizumab and Erlotinib

INTERVENTIONS:
Drug: Bevacizumab and Erlotinib — Bevacizumab administered intravenously at dose 10 mg/kg every 2 wks. Erlotinib administered orally, continuously once daily in fasting state for each 42-day cycle. Dose of erlotinib is based on prior erlotinib monotherapy trial in RMG. It will be 200 mg/day for pts not on cytochrome P450 3A4 (CYP3A4)-enzyme inducing anti-epileptic drugs & 500 mg/day for pts on EIAEDs.
  It is possible that taking erlotinib w regular medications or supplements may change how erlotinib, subject's regular medications, or subject's regular supplements work. Treatment will continue until either evidence of progressive disease, unacceptable toxicity, non-compliance w study follow-up, or withdrawal of consent.
  Other Names: Bevacizumab; Erlotitnib; Avastin; Tarceva

SUMMARY:
Primary objective:

To estimate 6-month progression free survival probability of pts w recurrent malignant gliomas treated w erlotinib + bevacizumab.

Secondary Objectives:

To evaluate safety & tolerability of erlotinib + bevacizumab among pts w recurrent malignant gliomas To evaluate radiographic response of pts w recurrent malignant gliomas treated w erlotinib + bevacizumab To evaluate pharmacokinetics of erlotinib when administered to pts w recurrent malignant gliomas; & to examine relationship of clinical response to Epidermal Growth Factor (EGFR) expression, amplification, & v-III mutation, phosphatase and tensin homolog (PTEN) expression, vascular endothelial growth factor (VEGF) expression, vascular endothelial growth factor receptor 2 (VEGFR-2) & phosphorylated protein kinase B (PKB/Akt) in archival tumor samples

DETAILED DESCRIPTION:
Exploratory, Phase II study designed to assess anti-tumor activity of combinatorial regimen consisting of erlotinib + bevacizumab among pts w recurrent malignant glioma. Signal transduction inhibitors, such as erlotinib, as well as anti-angiogenic agents, such as bevacizumab, are expected to exert a cytostatic anti-tumor effect. Primary endpoint of study is probability of progression-free survival at 6 months. An important secondary objective is to further assess the safety of erlotinib + bevacizumab for pts w RMG. Pharmacokinetic studies included in protocol will evaluate impact of enzyme-inducing anti-epileptic drugs (EIAEDs) on metabolism of erlotinib.

If study demonstrates that combo regimen of erlotinib + bevacizumab is associated w encouraging anti-tumor activity among pts w recurrent malignant glioma (RMG), further assessment of regimen in additional ph II & possibly ph III studies, will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Pts have histologically confirmed diagnosis of recurrent/progressive WHO gr III & IV MG & meet following inclusion criteria:
* Age >18 yrs
* Interval of >4 wks since prior surgery
* Interval of >4 wks since prior external beam radiation therapy (XRT) or chemo, unless there is unequivocal evidence of progressive disease & pts have recovered from all anticipated toxicity of most recent therapy
* Karnofsky performance status score >60
* Hematocrit > 29 percent, absolute neutrophil count (ANC) >1,500 cells/microliter, platelets >100,000 cells/microliter
* Serum creatinine <.5mg/dl, blood urea nitrogen (BUN) <25 mg/dl, serum glutamate oxaloacetate transaminase (SGOT) & bilirubin <1.5 x upper limit of normal (ULN)
* For pts on corticosteroids, they have been on stable dose for 1 wk prior to entry
* Pts have had prior bevacizumab are eligible however interval of >6 wks must have elapsed since their last dose
* Signed informed consent approved by Institutional Review Board (IRB) prior to patient entry;
* If sexually active, pts must agree to take contraceptive measures for duration of treatments

Exclusion Criteria:

* Prior therapy w either bevacizumab/EGFR-directed agents
* >3 prior recurrences
* Pregnancy/breast feeding
* Co-medication w immuno-suppressive agents other than corticosteroids including but not limited to cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil
* Evidence of central nervous system (CNS) hemorrhage on baseline MRI on CT scan
* Pts who require therapeutic anti-coagulation
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring IV antibiotics & psychiatric illness/social situations that would limit compliance w study requirements, or disorders associated w significant immunocompromised state
* Pts w another primary malignancy that has required treatment within past year
* Pts w acute/chronic renal insufficiency/those w acute renal insufficiency of any severity due to hepato-renal syndrome/in peri-operative liver transplantation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- [Derived] Sathornsumetee S, Desjardins A, Vredenburgh JJ, McLendon RE, Marcello J, Herndon JE, Mathe A, Hamilton M, Rich JN, Norfleet JA, Gururangan S, Friedman HS, Reardon DA. Phase II trial of bevacizumab and erlotinib in patients with recurrent malignant glioma. Neuro Oncol. 2010 Dec;12(12):1300-10. doi: 10.1093/neuonc/noq099. Epub 2010 Aug 17. PMID 20716591
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open for recruitment from February 2007 to May 2008. Subjects recruited in the Preston Robert Tisch Brian Tumor Center at Duke University Medical Center (DUMC).
Groups:
- WHO Grade III: WHO Grade III Malignant Glioma
  Bevacizumab administered intravenously at dose 10 mg/kg every 2 wks. Erlotinib administered orally, continuously once daily in fasting state for each 42-day cycle. It will be 200 mg/day for pts not on cytochrome P450 3A4 (CYP3A4)-enzyme inducing anti-epileptic drugs & 500 mg/day for pts on EIAEDs.
- WHO Grade IV: WHO Grade IV Malignant Glioma
  Bevacizumab administered intravenously at dose 10 mg/kg every 2 wks. Erlotinib administered orally, continuously once daily in fasting state for each 42-day cycle. It will be 200 mg/day for pts not on cytochrome P450 3A4 (CYP3A4)-enzyme inducing anti-epileptic drugs & 500 mg/day for pts on EIAEDs.
Period: Overall Study
Arm/Group | WHO Grade III | WHO Grade IV
Started | 32 | 25
Completed | 32 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Who Grade III: Who Grade III Malignant Glioma
- WHO Grade IV: WHO Grade IV Malignant Glioma
- Total: Total of all reporting groups
Arm/Group | Who Grade III | WHO Grade IV | Total
Number analyzed (Participants) | 32 | 25 | 57
Age Continuous [Median (Standard Deviation); unit: years] | 48.8 (12.8) [26.0 to 72.2] | 51.5 (13.4) [24.1 to 70.4] | 49.98 (13.05) [24.1 to 72.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 24 | 13 | 37

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-free Survival
Description: The proportion of patients alive and progression free at 6 months
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Who Grade III | WHO Grade IV
Number analyzed (Participants) | 32 | 25
proportion of participants | .438 [.265 to .598] | .292 [.130 to .476]

2. Secondary Outcome: Radiographic Response
Description: The number of participants with complete or partial response as determined by the following criteria:
  * Complete response (CR): Disappearance of all enhancing tumor on contrast enhanced MRI scan. Patient must be off steroids or only on adrenal maintenance doses.
  * Partial response (PR): Greater than or equal to a 50% reduction in the size (products of the largest perpendicular diameters) for all enhancing lesions. No new lesions may arise. Steroids must be stable or decreasing dose.
Time Frame: Patients were followed for the duration of the study, with a median follow-up of 103 weeks for grade III participants and 141.8 weeks for grade IV participants
Measure: Number; unit: participants
Arm/Group | Who Grade III | WHO Grade IV
Number analyzed (Participants) | 32 | 25
participants
  Complete | 1 | 1
  Partial | 9 | 11

3. Secondary Outcome: Pharmacokinetics of Erlotinib: Cmax
Description: Day 1 and Day 42 of Dosing Erlotinib in Cycle 1: Maximum Concentration (ng/mL) (Cmax) for subjects receiving 500 mg (Enzyme-Inducing Anti-epileptic Drug, EIAED) or 200 mg (non-EIAED) Erlotinib
Time Frame: Day 1 and 42 of Dosing Erlotinib
Population: 22 WHO Grade IV participants were available for pharmacokinetics studies of erlotinib
Measure: Median (Full Range); unit: ng/ml
Arm/Group | WHO Grade IV
Number analyzed (Participants) | 22
ng/ml
  Day1 Cmax{ng/ml}200mg n=12 | 794 [524 to 2200]
  Day1 Cmax{ng/ml}500mg n=10 | 1323 [317 to 2990]
  Day42 Cmax{ng/ml}200mg n=9 | 1320 [525 to 2940]
  Day42 Cmax{ng/ml}500mg n=9 | 1400 [716 to 3955]

4. Secondary Outcome: Pharmacokinetics of Erlotinib: AUC
Description: Day 1 and Day 42 of Dosing Erlotinib in Cycle 1: Area under the Curve (ng/mL.h) (AUC) for subjects receiving 500 mg (Enzyme-Inducing Anti-epileptic Drug, EIAED) or 200 mg (non-EIAED) Erlotinib
Time Frame: Day 1 and 42 of Dosing Erlotinib
Population: 22 WHO Grade IV participants were available for pharmacokinetics studies of erlotinib
Measure: Median (Full Range); unit: ng/ml.h
Arm/Group | WHO Grade IV
Number analyzed (Participants) | 22
ng/ml.h
  Day1 AUC 0-24{ng/ml.h} 200mg n=12 | 11072 [7850 to 30029]
  Day1 AUC 0-24{ng/ml.h} 500mg n=10 | 15611 [5295 to 40110]
  Day42 AUC 0-24{ng/ml.h}200mg n=9 | 26072 [8308 to 42878]
  Day42 AUC 0-24{ng/ml.h}500mg n=9 | 21421 [11680 to 55960]

5. Secondary Outcome: Association of Biomarkers and One-year Survival - Epidermal Growth Factor (EGFR)
Description: Archival tumor samples from grade IV participants were examined by immunohistochemistry for biomarkers.
Time Frame: 1 year
Population: Tumors from 22 GBM participants were available to undergo immunohistochemical staining to identify potential biomarkers of response or survival benefit. One tumor had an insufficient measurement for analysis
Measure: Number; unit: participants
Groups:
- Positive Expression: EGFR positive expression
- Negative Expression: EGFR negative expression
Arm/Group | Positive Expression | Negative Expression
Number analyzed (Participants) | 20 | 1
participants | 7 | 0
Statistical Analysis 1: Comparison: Positive Expression vs Negative Expression; Test type: Superiority or Other; p = 1.0, Fisher Exact

6. Secondary Outcome: Association of Biomarkers and One-year Survival - EGFR vIII
Description: Archival tumor samples from grade IV participants were examined by immunohistochemistry for biomarkers.
Time Frame: 1 year
Population: Tumors from 22 GBM participants were available to undergo immunohistochemical staining to identify potential biomarkers of response or survival benefit.
Measure: Number; unit: participants
Groups:
- Positive Expression: EGFR vIII positive expression
- Negative Expression: EGFR vIII negative expression
Arm/Group | Positive Expression | Negative Expression
Number analyzed (Participants) | 5 | 17
participants | 1 | 7
Statistical Analysis 1: Comparison: Positive Expression vs Negative Expression; Test type: Superiority or Other; p = .613, Fisher Exact

7. Secondary Outcome: Association of Biomarkers and One-year Survival - Phosphatase and Tensin Homologue (PTEN)
Description: Archival tumor samples from grade IV participants were examined by immunohistochemistry for biomarkers.
Time Frame: 1 year
Population: as for outcome 5
Measure: Number; unit: participants
Groups:
- Intact: PTEN Intact
- Loss: PTEN Loss
Arm/Group | Intact | Loss
Number analyzed (Participants) | 2 | 19
participants | 1 | 7
Statistical Analysis 1: Comparison: Intact vs Loss; Test type: Superiority or Other; p = 1.0, Fisher Exact

8. Secondary Outcome: Association of Biomarkers and One-year Survival - Phosphorylated Protein Kinase B (pAKT)
Description: Archival tumor samples from grade IV participants were examined by immunohistochemistry for biomarkers.
Time Frame: 1 year
Population: Tumors from 22 GBM participants were available to undergo immunohistochemical staining to identify potential biomarkers of response or survival benefit. Four tumors had an insufficient measurement for analysis.
Measure: Number; unit: participants
Groups:
- Positive Expression: pAKT positive expression
- Negative Expression: pAKT negative expression
Arm/Group | Positive Expression | Negative Expression
Number analyzed (Participants) | 16 | 2
participants | 6 | 1
Statistical Analysis 1: Comparison: Positive Expression vs Negative Expression; Test type: Superiority or Other; p = 1.0, Fisher Exact

9. Secondary Outcome: Association of Biomarkers and One-year Survival - Phosphorylated Mitogen-activated Protein Kinase (pMAPK)
Description: Archival tumor samples from grade IV participants were examined by immunohistochemistry for biomarkers.
Time Frame: 1 year
Population: Tumors from 22 GBM participants were available to undergo immunohistochemical staining to identify potential biomarkers of response or survival benefit. Six tumors had an insufficient measurement for analysis.
Measure: Number; unit: participants
Groups:
- Positive Expression: pMAPK positive expression
- Negative Expression: pMAPK negative expression
Arm/Group | Positive Expression | Negative Expression
Number analyzed (Participants) | 12 | 4
participants | 5 | 1
Statistical Analysis 1: Comparison: Positive Expression vs Negative Expression; Test type: Superiority or Other; p = 1.0, Fisher Exact

10. Secondary Outcome: Association of Biomarkers and One-year Survival - Vascular Endothelial Growth Factor (VEGF)
Description: Archival tumor samples from grade IV participants were examined by immunohistochemistry (IHC) for biomarkers. The IHC expression score is the product of the percentage of cancer cells positive for VEGF multiplied by the overall intensity of staining, ranging from 0 to 3+. This produces a score ranging from 0 to 300.
Time Frame: 1 year
Measure: Median (Full Range); unit: IHC Expression Score
Groups:
- Patients Who Survived At Least 1 Year: Patients who survived at least 1 year
- Patients Who Survived Less Than 1 Year: Patients who survived less than 1 year
Arm/Group | Patients Who Survived At Least 1 Year | Patients Who Survived Less Than 1 Year
Number analyzed (Participants) | 8 | 14
IHC Expression Score | 40 [4 to 120] | 60 [20 to 160]
Statistical Analysis 1: Comparison: Patients Who Survived At Least 1 Year vs Patients Who Survived Less Than 1 Year; Test type: Superiority or Other; p = .179, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Association of Biomarkers and One-year Survival - VEGFR-2
Description: Archival tumor samples from grade IV participants were examined by immunohistochemistry (IHC) for biomarkers. The IHC score is the product of the percentage of cancer cells positive for VEGFR-2 multiplied by the overall intensity of staining, ranging from 0 to 3+. This produces a score ranging from 0 to 300.
Time Frame: 1 year
Measure: Median (Full Range); unit: IHC Expression Score
Arm/Group | Patients Who Survived At Least 1 Year | Patients Who Survived Less Than 1 Year
Number analyzed (Participants) | 8 | 14
IHC Expression Score | 50 [20 to 100] | 120 [40 to 160]
Statistical Analysis 1: Comparison: Patients Who Survived At Least 1 Year vs Patients Who Survived Less Than 1 Year; Test type: Superiority or Other; p = .008, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: The length of time that the subjects were receiving treatment and then 30 days after treatment termination.
Description: Adverse events were collected using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0, but were converted to CTCAE version 4.0 for entry into ClinicalTrials.gov
Groups:
- All Patients: All Patients
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 20/57
Other Adverse Events (participants affected / at risk) | 52/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=57)
Colonic ulcer (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Death NOS (General disorders) | 2
Edema limbs (General disorders) | 1
Gait disturbance (General disorders) | 1
Device related infection (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Wound dihiscence (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Intracranial hemorrhage (Nervous system disorders) | 2
Ischemia cerebrovascular (Nervous system disorders) | 1
Nervous system disorders-Other, specify: Visual Hallucinations (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Personality change (Psychiatric disorders) | 1
Psychosis (Psychiatric disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Thromboembolic event (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=57)
Anemia (Blood and lymphatic system disorders) | 10
Blurred vision (Eye disorders) | 14
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 28
Mucositis oral (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 5
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 40
Fever (General disorders) | 3
Skin infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 5
Alanine aminotransferase increased (Investigations) | 10
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 6
Investigations-Other, specify: Total protein, low (Investigations) | 15
Platelet count decreased (Investigations) | 6
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 23
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
Hypocalcemia (Metabolism and nutrition disorders) | 10
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Ataxia (Nervous system disorders) | 17
Cognitive disturbance (Nervous system disorders) | 20
Dizziness (Nervous system disorders) | 17
Dysphasia (Nervous system disorders) | 13
Headache (Nervous system disorders) | 20
Memory impairment (Nervous system disorders) | 25
Nervous system disorders-Other, specify: Mood Alteration, NOS (Nervous system disorders) | 8
Peripheral motor neuropathy (Nervous system disorders) | 26
Peripheral sensory neuropathy (Nervous system disorders) | 15
Pyramidal tract syndrome (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 13
Tremor (Nervous system disorders) | 14
Agitation (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 14
Confusion (Psychiatric disorders) | 20
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 24
Libido decreased (Psychiatric disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 5
Reproductive system and breast disorders-Other, specify: Sexual Dysfunction (Reproductive system and breast disorders) | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 44
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes